CLINICAL TRIAL: NCT04862390
Title: Incidence of Hypoglycemia in Pregnant Women With or Without Diabetes During Fasting in Ramadan
Brief Title: Incidence of Hypoglycemia in Pregnant Ladies With or Without Gestational Diabetes Fasting Ramadan
Status: Completed | Type: Observational
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: NRJ21J/034/02
Record Dates: First submitted 2021-04-25; First posted 2021-04-28 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy in Diabetic
Keywords: Pregnant, gestational diabetes, fasting
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes, Gestational; Fasting | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Pregnancy: Pregnant women with no diabetes
  Interventions: Device: Continuous glucose monitoring
- Gestational diabetes on diet alone
  Interventions: Device: Continuous glucose monitoring
- Gestational diabetes on diet + Metformin therapy
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Home continuous glucose monitoring to be installed for two weeks during fasting Ramadan

SUMMARY:
The physiological change in food and sleep pattern during Ramadan impacted hypoglycemia risks among pregnant women. Few studies investigated the incidence of hypoglycemia pregnant women with or without diabetes during fasting in Ramadan in Saudi Arabia. This study aims to understand the glucose variability in pregnant women during fasting Ramadan in Saudi Arabia.

DETAILED DESCRIPTION:
Women with normal pregnancy will be compared to women with gestational diabetes on diet or Metformin alone during Fasting Ramadan. They will be monitored and will be observed for incidence of hypoglycemia using continuous glucose monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. Pregnant women without diabetes.
3. Pregnant women with diabetes (pregestational and gestational) on diet +/- metformin.
4. Dedicated to applying a continuous glucose monitoring (CGM) device.

Exclusion Criteria:

1. Age below18 years
2. Pregnant women with diabetes on insulin (type 1 and type 2 diabetes)
3. Renal and liver impairment.
4. Adrenal insufficiency
5. Psychiatric diseases.

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant ladies without gestational diabetes (GDM) and with GDM on diet or metformin attending the endocrine and obstetric clinics at National Guards Hospital Jeddah, and who intend to fast Ramadan will be recruited over 2 months period prior to Ramadan. Those who accept and fulfill the inclusion criteria will be consented to participate. During Ramadan they will be requested to do home glucose monitoring which is part of standard of care and will also be put on glucose sensors for 14 days, after which reprots will be downloaded
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia incidence with fasting | 1 month
  To estimate the incidence of hypoglycemia defined as blood glucose < 70 mg/dl during fasting in pregnant women with gestational diabetes on diet therapy or metformin alone compared to women without diabetes

SECONDARY OUTCOMES:
Glucose variability during fasting Ramadan | 1 month
  To estimate the difference in the groups in glucose variability
Number of days that needed to break fasting | 1 month
  To estimate the difference in the groups in number of days that needed to break fasting
Time in range (TIR) | 1 month
  TIR is defined as blood glucose range between 63-140 mg/dl (3.5-7.8 mmol/L) according to ADA guideline.
Time above range (TAR) | 1 month
  TAR that defined as blood glucose range >140 mg/dl (>7.8 mmol/L) according to ADA guideline.
Time below range (TBR) | 1 month
  TBR that defined as blood glucose range < 60 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Reem M Alamoudi, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- KingAbullahIMRC, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided